CLINICAL TRIAL: NCT00792480
Title: Does Dietary and Lifestyle Counseling Prevent Excessive Weight Gain During Pregnancy? A Randomized Controlled Trial
Acronym: WIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resident research project limited by restrictions of residency program.
Sponsor: Carolinas Medical Center (Other)
Responsible Party: Shelly Asbee, MD, PI, Lake Norman Ob/Gyn
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WIP 06-05-04A
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-11

CONDITIONS: Obesity; Pregnancy
Keywords: Obesity; Pregnancy; Exercise; Nutrition; obesity in pregnancy
MeSH Terms: conditions — Obesity; Motor Activity; Pregnancy in Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Counseling Group (Experimental)
  Interventions: Behavioral: Dietary and lifestyle counseling
- Routine care group (No Intervention): The routine care group took part in an initial physical exam and history, routine labs, and routine visits per American College of Obstetrics & Gynecology (ACOG) standards. The only counseling on diet and exercise during pregnancy was that included in our standard prenatal booklet "What to do When You're Having a Baby" by Gloria Mayer (Institute for Health Advancement, 2003, La Habra, CA). At each routine obstetric appointment, the participant's weight was measured recorded in the medical chart. The healthcare provider did not counsel the participant regarding any changes in diet or lifestyle.

INTERVENTIONS:
Behavioral: Dietary and lifestyle counseling — The intervention group will undergo a complete history and physical with attention to prepregnancy weight, current weight, height, and BMI. At the initial visit, they will meet with a registered dietician to receive a standardized counseling session, including information on pregnancy-specific dietary and lifestyle choices. The patient will be instructed to engage in moderate intensity exercise at least 3 times per week and preferably 5 times per week. They will also receive information on the appropriate weight gain during pregnancy using the IOM guidelines. Each subject will meet with the dietician only at the time of enrollment.
  At each routine obstetric appointment, the participant's weight will be measured and charted on an IOM Gestational Weight Gain Grid in front of the participant. The healthcare provider will inform the participant if her weight gain was at the appropriate level and counsel her accordingly regarding increasing or decreasing her intake and exercise.
  Arms: Intensive Counseling Group

SUMMARY:
The purpose of this study is to determine if an organized, consistent program of dietary and lifestyle counseling will prevent excessive gestational weight gain.

DETAILED DESCRIPTION:
Excessive gestational weight gain is common with about one third of women gaining more weight in pregnancy than is recommended. Unfortunately, the prevalence of excessive gestational weight gain is increasing. Gestational weight gain greater than that recommended by the Institute of Medicine (IOM) is associated with increased risk of gestational complications (hypertension, diabetes, and preeclampsia), infant macrosomia, and complications in delivery including increased risk of cesarean delivery. Currently, there is no evidence-based prenatal counseling protocol available to prevent excessive gestational weight gain. We hypothesize that consistent counseling on appropriate pregnancy diet, weight gain, and the potential complications of excessive gestational weight gain will result in fewer women gaining above the IOM recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Establish prenatal care at 6 - 16 weeks gestation
2. 18-49 years of age
3. Receive their entire prenatal care at the Resident Obstetrics Clinic
4. English and/or Spanish speaking
5. Singleton gestation.

Exclusion Criteria:

1. Establish prenatal care >16 weeks gestation
2. Non-English or non-Spanish speaking
3. Multiple gestation pregnancy
4. BMI > 40
5. Preexisting diabetes, untreated thyroid disease, or hypertension requiring medication or other medical conditions that might affect body weight
6. Delivery at institution other than CMC-Main
7. Pregnancy ending in a premature delivery (< 37 weeks)
8. Limited prenatal care (<4 visits)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2005-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The investigators primary outcome is the rate of adherence to the IOM guidelines between our study groups. | 3 - 6 months

SECONDARY OUTCOMES:
The investigators secondary outcomes will include the effect of weight gain on mode of delivery, rate of operative vaginal delivery, infant weight, and the incidence of preeclampsia, GDM, vaginal/perineal lacerations, and shoulder dystocia. | 3 - 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shelly M Asbee, M.D., Principal Investigator — Lake Norman Ob/Gyn
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

REFERENCES:
- [Derived] Asbee SM, Jenkins TR, Butler JR, White J, Elliot M, Rutledge A. Preventing excessive weight gain during pregnancy through dietary and lifestyle counseling: a randomized controlled trial. Obstet Gynecol. 2009 Feb;113(2 Pt 1):305-12. doi: 10.1097/AOG.0b013e318195baef. PMID 19155899